CLINICAL TRIAL: NCT02297347
Title: The Brain, Neurological Features and Neuropsychological Functioning in Adults With Sapropterin Dihydrochloride Treated Phenylketonuria
Brief Title: The Brain and Neuropsychological Functioning in Adults With Sapropterin Dihydrochloride Treated Phenylketonuria
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Susan Waisbren, Associate Professor of Psychology, Boston Children's Hospital
Other Study IDs: IRB-P00015326
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Phenylketonuria
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Newborn screening and early treatment prevent the most severe manifestations of phenylketonuria (PKU). However, executive functioning deficits, attention deficit disorder, slow processing speed, and visual-motor problems commonly occur. Many adults with this disorder also suffer depression and anxiety. In this study the investigators will examine adults with PKU on sapropterin dihydrochloride (Kuvan) treatment for PKU and compare their results to those of subjects with PKU not on Kuvan. Using magnetic resonance imaging (MRI) techniques, including novel MR spectroscopy (MRS) the investigators hope to discover why this distinct constellation of deficits occurs in PKU. Adult subjects with PKU will undergo a comprehensive MRI evaluations, including a novel method of MR spectroscopy to determine brain phenylalanine levels. In addition, participants will receive neurological and neuropsychological examinations and dietary evaluation.

DETAILED DESCRIPTION:
Phenylketonuria (PKU, OMIM 261600), an autosomal recessive disorder, affects approximately 1:11,000 individuals in the United States. In PKU, mutations in the gene responsible for the liver enzyme phenylalanine hydroxylase (PAH) result in reduced or absent conversion of phenylalanine (Phe) to tyrosine (Tyr) and subsequently to elevated plasma concentrations of Phe and reduced concentrations of Tyr (Scriver and Kaufman, 2001). Untreated PKU results in progressive, neurological decline by 6-12 months of age (Koch et al, 1971). Even with early detection and treatment with a Phe-restricted diet, patients experience neurocognitive deficits (Waisbren et al, 1994) and psychiatric disturbances as they get older (Brumm et al, 2010; Bilder et al, 2013; Weglage et al, 2013) as well as white matter abnormalities detected through magnetic resonance imaging (MRI) (Mastrangelo et al, 2015).

In treated PKU, neuropsychological functioning is associated with exposure to elevated blood phenylalanine levels (Jahja et a;. 2017; and decreased blood tyrosine (Luciana, Sullivan, Nelson, 2001). However, the extent to which these biomarkers confer risks to cognitive and emotional well-being varies dramatically, with some individuals experiencing serious deficits and others functioning normally despite equally high phenylalanine or depleted tyrosine levels in blood (Rajabi, Waisbren and Levy, 2016; Manti et al, 2017 ). One explanation is that blood Phe and Tyr do not represent exposure in the brain (Diamond et al, 1997; Surtees and Blau, 2000).

Previously, we reported on an improved method for measuring brain Phe and brain Tyr in PKU (Waisbren et al, 2016) using two dimensional shift correlated magnetic resonance spectroscopy (COSY) (Thomas et al, 2001). This allows for the unambiguous identification of cerebral metabolites that could not be detected using conventional MRS methods due to spectral overlap. By obtaining multiple acquisitions at different echo times, a second chemical shift domain allows for metabolites to be identified by two chemical shifts instead of just one based on scalar coupling of different proton groups. The concentration of the metabolite is therefore shown in the third dimension. By visualizing the COSY data in three dimensions, smaller resonances that would have been obscured by larger resonances can be measured (Figure 1). Different brain regions, separating white and gray matter tissue, can be assessed with this method as a smaller voxel can be used.

In our previous study, we demonstrated that COSY could be used to quantify brain Phe and brain Tyr in two brain regions in adults with treated PKU without the need for a phenylalanine load. We also examined the relationship between these biomarkers and neuropsychological functioning and found that associations were in the expected direction, with higher brain Phe and lower brain Tyr related to poorer functioning (Waisbren et al, 2016).

The aims of the study reported here were to examine the relationships between blood and brain concentrations of Phe and Tyr in patients on sapropterin dihydrochloride (BH4 or Kuvan) and to assess the relationships between these biomarkers and neuropsychological functioning.

ELIGIBILITY:
Inclusion Criteria:

* Adult with classic PKU currently on Kuvan treatment for at least one month.
* Age 18-55 years
* Medical Records available that include blood phenylalanine levels during the first 6 years of life.
* Capable of providing informed consent
* Able to undergo MRI procedures without sedating medication
* Does not have metal implants, braces, or permanent retainers.

Exclusion Criteria:

* Mild PKU or mild hyperphenylalaninemia
* Less than 18 years old or greater than 55 years old
* No medical records available for the first 6 years of life
* Not capable of providing informed consent
* Not able to undergo MRI without sedating medication
* Has metal implants, braces or permanent retainers
* Currently involved in any clinical trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults with PKU on Kuvan treatment for at least one month prior to enrolling in the study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Phenylalanine (phe) level in the brain as determined by MR Spectroscopy | one day
  Brain phe described as umol/L through MR Spectroscopy in both the , posterior cingulate gyrus (PCG) and parietal white matter (PWM)

SECONDARY OUTCOMES:
Full Scale IQ | one day
  Full Scale IQ is obtained from the Wechsler Abbreviated Scale of Intelligence
Brain tyrosine (tyr) level as determined by MR Spectroscopy | one day
  Brain tyr described as umol/L through MR Spectroscopy in both the , posterior cingulate gyrus (PCG) and parietal white matter (PWM)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E. Waisbren, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States